CLINICAL TRIAL: NCT05337111
Title: Differences in Cardiorespiratory Fitness and Fat Oxidation at Rest and During Exercise in Chinese, Indian and Malay Men With Elevated Body Mass Index.
Brief Title: Fitness and Fat Oxidation in Overweight Chinese, Indian and Malay Men
Status: Completed | Type: Observational
Sponsor: Nanyang Technological University (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Other Study IDs: 2017-T1-002-036
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chinese men: Chinese men based on self-identity for three generations (parents and grandparents), age 25 - <45 years, who are physically inactive (< 150 minutes moderate or < 75 minutes vigorous leisure-time physical activity per week), with elevated body mass index (>23-<30 kg/m2) for Asians. Single measure of CRF, resting fat oxidation and fat oxidation during graded exercise.
  Interventions: Other: Cardiorespiratory fitness test; Other: Resting measure of fat oxidation; Other: Maximum fat oxidation test
- Indian men: Indian men based on self-identity for three generations (parents and grandparents), age 25 - <45 years, who are physically inactive (< 150 minutes moderate or < 75 minutes vigorous leisure-time physical activity per week), with elevated body mass index (>23-<30 kg/m2) for Asians. Single measure of CRF, resting fat oxidation and fat oxidation during graded exercise.
  Interventions: Other: Cardiorespiratory fitness test; Other: Resting measure of fat oxidation; Other: Maximum fat oxidation test
- Malay men: Malay men based on self-identity for three generations (parents and grandparents), age 25 - <45 years, who are physically inactive (< 150 minutes moderate or < 75 minutes vigorous leisure-time physical activity per week), with elevated body mass index (>23-<30 kg/m2) for Asians. Single measure of CRF, resting fat oxidation and fat oxidation during graded exercise.
  Interventions: Other: Cardiorespiratory fitness test; Other: Resting measure of fat oxidation; Other: Maximum fat oxidation test

INTERVENTIONS:
Other: Cardiorespiratory fitness test — Progressive submaximal exercise test on a treadmill to predict cardiorespiratory fitness
  Other Names: Graded exercise test, submaximal oxygen uptake test
Other: Resting measure of fat oxidation — Use of ventilated hood attached to automated metabolic cart to measure substrate oxidation at rest
  Other Names: Resting energy expenditure, resting substrate oxidation test
Other: Maximum fat oxidation test — Progressive exercise test to determine maximum fat oxidation during exercise

SUMMARY:
South Asian men have lower cardiorespiratory fitness (CRF) than white men which is associated with a reduced capacity to oxidise fat during exercise. This is a risk factor for weight gain/regain. Whilst comparisons with Europeans are valuable, Asians are not a homogenous group and substantial differences in obesity and body fat partitioning exist with ethnicity. This cross-sectional pilot investigation aims to compare CRF and fat oxidation at rest and during exercise in Chinese, Indian and Malay men (from Singapore) with elevated BMI (23 -30 kg/m2). Forty-five men (15 each ethnicity) with elevated body mass index (23 -30 kg/m2) will complete testing in a fasted state on two separate mornings separated by ≥72 hours: (i) for a measure of CRF; and (ii) for a measure of fat oxidation at rest and during incremental exercise.

DETAILED DESCRIPTION:
South Asian men have lower cardiorespiratory fitness (CRF) than white men which is associated with a reduced capacity to oxidise fat during exercise. This is a risk factor for weight gain/regain. Whilst comparisons with Europeans are valuable, Asians are not a homogenous group and substantial differences in obesity and body fat partitioning exist with ethnicity. This cross-sectional pilot investigation aims to compare CRF and fat oxidation at rest and during exercise in Chinese, Indian and Malay men (from Singapore) with elevated BMI (23 -30 kg/m2). Forty-five men (15 each ethnicity) with elevated body mass index (23 -30 kg/m2) will complete testing in a fasted state on two separate mornings separated by ≥72 hours: (i) for a measure of CRF; and (ii) for a measure of fat oxidation at rest and during incremental exercise. A submaximal exercise test will be used to estimate CRF (maximum oxygen uptake, VO2max) during walking using a standard protocol where subjects walk on a treadmill at 5 km/h with regular increments in gradient until individuals reach 80% of their estimated maximum heart rate [220 - age (years)]. Perceived exertion will be monitored assessed periodically during the test and expired gases continuously measured via a mouthpiece attached to an automated metabolic cart (Parvomedics MMS-2400; Parvomedics, Sandy, UT). Oxygen consumption will be extrapolated to estimate VO2max based on estimated maximum heart rate. Resting fat oxidation will be determined via a 30 minute measure of expired gases under a ventilated hood attached to an automated metabolic cart. Fat oxidation during exercise will be determined via walking on a treadmill with increments in speed and gradient until the respiratory exchange ratio is ≥ 0.95. Primary outcomes will be compared among groups and adjusted for any covariates (e.g., BMI, body fat percentage) as necessary.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 25 - <45 years
* Chinese, Indian or Malay based on self-identity for three generations (parents and grandparents)
* BMI ≥ 23 - < 30 kg/m2 and/or waist circumference ≥ 90 cm
* physically inactive defined as < 150 minutes moderate or < 75 minutes vigorous leisure-time physical activity per week, or the equivalent combination of both

Exclusion Criteria:

* females
* personal history of cardio-metabolic diseases
* dieting (i.e. restricting food/energy intake)
* smokers
* consuming alcohol > 3 times per week with > 3 drinks per time
* using any medications which affect carbohydrate or lipid metabolism
* any lower body injuries
* fasting blood glucose > 6.1 mmol/L

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy but physically inactive Chinese, Indian and Malay men aged 21-45 years with an elevated body mass index for Asians.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 1 day (Single measurement)
  Predicted measure of maximum oxygen uptake during exercise
Resting fat oxidation | 1 day (Single measurement)
  Measure of amount of fat oxidised whilst at rest in the postabsorptive (fasting) state
Maximum fat oxidation (exercise) | 1 day (Single measurement)
  Measure of maximum amount of fat oxidised whilst exercising in the postabsorptive state

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F Burns, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
A copy of the anonymised data relating to this study will be made available in the Data Repository of the National Institute of Education (Singapore) after publication. Access to the data will be via reasonable request to the Principal Investigator.

REFERENCES:
- [Derived] Demashkieh M, Dalan R, Burns SF. Cardiorespiratory fitness and fat oxidation during exercise in Chinese, Indian, and Malay men with elevated body mass index. Appl Physiol Nutr Metab. 2022 Aug 1;47(8):888-892. doi: 10.1139/apnm-2022-0106. Epub 2022 Jun 9. PMID 35679614